CLINICAL TRIAL: NCT03770117
Title: A Pilot Study of the Effect of Prehabilitation on Markers of Sarcopenia in Patients Undergoing Pancreatoduodenectomy for Malignant Disease
Brief Title: Study of the Effect of Prehabilitation on Markers of Sarcopenia in Patients Undergoing Pancreatoduodenectomy for Malignant Disease
Acronym: SIPUP
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00101
Record Dates: First submitted 2018-12-07; First posted 2018-12-10 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreas; Cancer; Sarcopenia; Cachexia; Prehabilitation; Pancreatoduodenectomy
MeSH Terms: conditions — Neoplasms; Sarcopenia; Cachexia | interventions — Preoperative Exercise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prehabilitation: In this arm of the study, participants will undergo prehabilitation prior to surgery. This is intended to increase the participants overall health prior to surgery to try and increase their general well-being during and after surgery.
  Prehabilitation is multimodal therapy comprising:
  1. Assessment for malnutrition and nutritional support dependent on the outcome
  2. Optimisation of management of pancreatic exocrine insufficiency
  3. Assessment of muscle mass and strength
  4. Individually tailored, goal directed exercise regimen under the care of physiotherapy
  Interventions: Procedure: Prehabilitation
- Standard Procedure: In this arm, participants will not receive any Rehabilitation prior to the surgery. This is the current standard care and will act as the control data for this study.
  Interventions: Procedure: Standard Procedure

INTERVENTIONS:
Procedure: Prehabilitation — Participants who underwent Prehabilitation will have their CT scans analysed.
  Groups: Prehabilitation
Procedure: Standard Procedure — Patients who underwent a panctratoduodenectomy and did not receive any Prehabilitation will have their CT scans analysed and compared.
  Groups: Standard Procedure

SUMMARY:
The aim of this study is to assess whether prehabilitation supervised by an appropriate multimodality team improves indices of sarcopenia in patients scheduled to undergo pancreatoduodenectomy.

DETAILED DESCRIPTION:
Cachexia is a hallmark feature of pancreatic cancer. Patients with features of cachexia have worse clinical outcomes. This includes a reduction in quality of life, reduced tolerance of therapy and a poorer prognosis . Specifically related to patients undergoing pancreatic surgery clinical evidence of cachexia is associated with higher perioperative complication rates. Sarcopenia, defined as a decreased muscle mass independent of fat mass, is a feature of the cachexia associated with pancreatic cancer. Patients with sarcopenia have progressive and generalised reduced muscle mass and function In patients undergoing surgery for pancreatic cancer sarcopenia has been associated with increased rates of complication and worse survival . Treatment of sarcopenia is difficult but includes nutritional support and pancreatic enzyme replacement therapy (PERT) aimed at reducing malabsorption. Whether measures aimed at combating sarcopenia can improve clinical outcomes following pancreatic surgery is currently unknown.

Prehabilitation is a multimodal therapeutic regimen aimed at improving the overall physical condition of patients prior to surgery with the intention of reducing the incidence of perioperative complications. Emerging evidence suggests that exercise prior to surgery for high risk patients scheduled to undergo major abdominal surgery improves aerobic capacity and can reduce the incidence of perioperative complications . The impact of prehabilitation undertaken prior to pancreatic surgery on perioperative complication rates has not yet been investigated.

The aim of this study is to assess whether prehabilitation supervised by an appropriate multimodality team improves indices of sarcopenia in patients scheduled to undergo pancreatoduodenectomy.

ELIGIBILITY:
Inclusion criteria

1. Patients treated by pancreatic resection
2. Surgery for malignancy
3. Patients aged over 16
4. CT scans available for assessment

Exclusion criteria

1. Patients scheduled for fast-track pancreatic resection as part of the jaundice pathway
2. Aged under 16
3. Patients not undergoing pancreatic resection

Ages: 16 Years to 100 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients who have had a pancreatoduodenectomy. Control group will have had standard care and these CT Scan results will be compared with those who have undergone prehabilitation.
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2018-10-04 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
CT Scan Comparison | Within last 5 years.
  CT Scans from patients which underwent the Prehabilitation & standard care will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Saurabh Jamdar, Study Chair — Manchester University NHS Foundation Trust
Locations (1):
- Manchester University NHS Foundation Trust, Manchester, Gtr Manchester, United Kingdom